CLINICAL TRIAL: NCT03248609
Title: Investigation of the Glycemic Index of Table Grape Varietals
Brief Title: Glycemic Index of Table Grape Varietals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1086796
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Milano grapes (Experimental): Unique grape varietal to test glycemic response.
  Interventions: Other: Milano grapes
- Table grapes (Active Comparator): Common grape varietal to test glycemic response and compare to the glycemic response elicited by the Milano grape varietal.
  Interventions: Other: Table grapes
- Grape juice (Active Comparator): Used to test the glycemic response without a complex food matrix and compare to the glycemic response elicited by the Milano grape varietal.
  Interventions: Other: Grape juice
- Glucose beverage (Placebo Comparator): Used to test the glycemic response with a standardized glucose beverage and compare to the glycemic response elicited by the Milano grape varietal.
  Interventions: Other: Glucose beverage

INTERVENTIONS:
Other: Milano grapes — Milano grapes to test post-prandial glycemic response
  Arms: Milano grapes
Other: Table grapes — Table grapes to test post-prandial glycemic response
  Arms: Table grapes
Other: Grape juice — Grape juice to test post-prandial glycemic response
  Arms: Grape juice
Other: Glucose beverage — Standardized glucose beverage to test post-prandial glycemic response
  Arms: Glucose beverage

SUMMARY:
Investigate the postprandial glycemic responses of healthy individuals when consuming commercially available table grape varietals or grape juice, compared to a standard amount of glucose.

DETAILED DESCRIPTION:
The study aims to investigate the postprandial glycemic responses of healthy individuals when consuming commercially available table grape varietals, compared to a standard amount of glucose. The study also aims to evaluate a new grape varietal, compared to other common table grapes, with regard to glycemic index and metabolic response related to inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 21-75 years of age
* BMI range 20-35

Exclusion Criteria:

* adults unable to consent, individuals who are not yet adults (children), pregnant women, and prisoners.
* BMI of >35 or morbid obesity.
* Diagnosed type 1 or 2 diabetes, fasting blood glucose of >125 mg/dl, or reported use of medications or supplements known to affect glucose metabolism (insulin, sulfonylureas, metformin, glucosidase inhibitors, thiazolidinedione, insulin sensitizers, GLP-1 mimetics).
* Medications known to affect gastrointestinal motility (prokinetic agents such as reglan).
* Renal, liver, pancreatic or cardiovascular disease, uncontrolled hypertension of > 160/90, inflammatory bowel disease, disorders of esophageal and gastrointestinal motility, previous gastric resection or restriction procedures, autoimmune or immunologic disorders, anemia, breastfeeding women
* Food allergy to grapes, or inability to tolerate gluten (celiac disease).
* Poor venous access.
* Smoking, illicit drug use, consuming >7 alcoholic drinks per week.
* Weight gain or loss of > 5 kg within the prior 6 months.
* Unwillingness to adhere to study protocol.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Glycemic Index | 3 hours
  The post-prandial glucose and insulin responses in healthy individuals to glucose containing foods or beverages.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis (Academic Surge, Ragle Human Nutrition Research Facility), Davis, California, United States

IPD SHARING:
Plan to Share IPD: No